CLINICAL TRIAL: NCT06372899
Title: Alternative Nicotine Delivery Systems as Potential Harm Reduction Tools for Persistent Cigarette Smokers
Brief Title: Noncombustible Nicotine Delivery Systems as Potential Harm Reduction Tools for Persistent Cigarette Smokers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Janet E. Audrain-McGovern, PhD, Professor, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UPCC 02024; R01CA290541-01A1 (NIH); 855140 (Other: University of Pennsylvania IRB Protocol Number)
Record Dates: First submitted 2024-04-12; First posted 2024-04-18 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: E-cigarette Use; Cigarette Smoking; Harm Reduction; Tobacco Use
MeSH Terms: conditions — Vaping; Cigarette Smoking; Harm Reduction; Tobacco Use | interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ECIGS (Experimental): Participants randomized to ECIGS will be provided with an e-cigarette device and be instructed to switch from smoking combustible cigarettes to using only the study-provided e-cigarette device. Participants will be able to choose between Tobacco, Menthol, Watermelon, and Blueberry flavored nicotine pods. They will receive their supply of nicotine pods in 7-day increments, based on baseline smoking behavior.
  Interventions: Other: E-cigarettes
- ONPS (Experimental): Participants randomized to ONPS will be provided with oral nicotine pouches and be instructed to switch from smoking combustible cigarettes to using only the study-provided nicotine pouches. Participants will be able to choose between Original, Mint, Berry, and Citrus flavored nicotine pouches. They will receive their supply of nicotine pouches in 7-day increments, based on baseline smoking behavior.
  Interventions: Other: Oral nicotine pouches

INTERVENTIONS:
Other: E-cigarettes — Participants randomized to ECIGS are instructed to switch from smoking combustible cigarettes to using e-cigarettes for 6 weeks. They will be provided with an e-cigarette device and nicotine pods.
  Arms: ECIGS
Other: Oral nicotine pouches — Participants randomized to ONPS are instructed to switch from smoking combustible cigarettes to using nicotine pouches for 6 weeks. They will be provided with nicotine pouches.
  Arms: ONPS

SUMMARY:
This between-subjects study aims to evaluate whether e-cigarettes (ECIGS) versus oral nicotine pouches (ONPS) more readily substitute for combustible cigarettes among 200 cigarette smokers. After measuring baseline cigarette smoking rate, participants will be randomized to ECIGS or ONPS and be instructed to switch (versus smoking cigarettes) over a 6-week period. Relative reductions in biomarkers of exposure will be measured. ECIG- and ONP-associated subjective reward and the reinforcing value of ECIGS and ONPS relative to combustible cigarettes will be assessed as mechanisms.

DETAILED DESCRIPTION:
E-cigarettes (ECIGS), and oral nicotine pouches (ONPs), expose users to few of the chemicals found in cigarette smoke and are thus promising noncombustible harm reduction tools for smokers who would not otherwise quit smoking. For their harm reduction potential to be realized, fundamental questions must be answered. One, can persistent smokers switch from combustible cigarettes to either ECIGS or ONPS? Two, what factors influence switching? Three, does one of these noncombustible alternatives expose users to lower levels of harmful chemicals than the other? The proposed research will fill these gaps in the evidence base by randomizing 200 persistent cigarette smokers to a six-week regimen of ECIGS or ONPS. Baseline smoking rate will be established during days 1-5. After biochemically confirmed overnight smoking abstinence, laboratory visits on days 6 and 7 will assess ECIG and ONP-associated subjective reward and the reinforcing value of either ECIGS or ONPS relative to combustible cigarettes. Participants will switch from cigarette smoking to ECIGS or ONPS for the following six weeks. The primary outcome measure is the longitudinal daily count of cigarettes from baseline to the end of the six-week switch period, measured via a validated collection protocol with cigarettes per day (cpd) at a 6-month follow-up as a secondary endpoint. Changes in biomarkers of potential harm, assessed at baseline and the end of the six-week switch phase, will be secondary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

1. Able to communicate fluently in English (i.e. speaking, writing, and reading)
2. Male and female smokers who are > 21 years of age and self-report smoking at least 5 cigarettes (menthol and/or non-menthol) per day for at least the last 6 months.
3. 5 or more failed quit attempts and the use of smoking cessation medication on at least one prior attempt.
4. Have a carbon monoxide (CO) greater than 10 ppm.
5. Not using any forms of nicotine regularly other than cigarettes
6. Be willing to switch to e-cigarettes or nicotine pouches for 6 weeks.
7. Plan to live in the area for the duration of the study.
8. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the combined consent and HIPAA form.

Exclusion Criteria:

Smoking Behavior

1. Regular use of nicotine-containing products other than cigarettes (e.g., chewing tobacco, snuff, snus, cigars, e-cigs, etc.). Regular e-cigarette and nicotine pouch use is defined as greater than 5 days/past 30 days.

   a. Participants agreeing to abstain from using nicotine-containing products other than cigarettes for the duration of the study will be considered eligible.
2. Current enrollment or plans to enroll in a smoking cessation program over the duration of the study.
3. Current use of smoking cessation medication
4. Provide a CO breath test reading less than 10 ppm at Intake.

Alcohol and Drug

1. History of substance abuse (other than nicotine dependence) in the past 12 months.
2. Current alcohol consumption that exceeds 20 standard drinks/week.
3. Current use of recreational drugs (other than nicotine and cannabis)
4. Breath alcohol reading (BrAC) greater than .000 at Intake.

Medical

1. Women, including all individuals assigned as "female" at birth, who are pregnant, breastfeeding, or planning a pregnancy over the duration of the study period.
2. Serious or unstable disease within the past year (e.g. cancer, heart disease). Applicable conditions will be evaluated on a case-by-case basis by the Principal Investigator.

Psychiatric

1. Lifetime history of schizophrenia or psychosis.

General Exclusion

1. Past, current, anticipated, or pending enrollment in another research program over the study period that could potentially impact subject safety, study data, and/or the study design as determined by the Principal Investigator.
2. Any medical condition, illness, disorder, adverse event (AE), or concomitant medication that could compromise participant safety or significantly impact study performance as determined by the Principal Investigator. Subjects may be deemed ineligible for any of the aforementioned reasons at any point throughout the study, as well as during the initial telephone screen.
3. Significant non-compliance with protocol and/or study design as determined by the Principal Investigator. Subjects may be deemed ineligible at any point throughout the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Cigarette Consumption | 42 days (days 8 - 49)
  The primary outcome is the longitudinal daily count of cigarettes from baseline to the end of the switch phase. Daily cigarette consumption will be determined by counting the daily spent cigarette filters returned for each of the 42 days (days 8 - 49).
Cigarette Smoking Across Follow-Up | 19 Weeks (Day 50-6-Month Follow-Up)
  Average cigarettes per day at the 6-month follow-up is a secondary endpoint, measured by the valid and reliable timeline follow-back (TLFB) interview.

SECONDARY OUTCOMES:
Biomarkers of Exposure: Carbon Monoxide (CO) | 49 days (days 1-49)
  Carbon Monoxide (CO) will be measured using a CO monitor. A CO > 5 ppm indicates combustible cigarette smoking.
Biomarkers of Exposure: Mean mid-expiratory forced expiratory flow (FEF25% - 75%) | 49 days (days 1-49)
  The mean mid-expiratory forced expiratory flow (FEF25% - 75%) is a measure of lung function and inflammation. FEF25% - 75% will be assessed using spirometry according to the American Thoracic Guidelines.
Biomarkers of Exposure: 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol (NNAL) | 49 days (days 1-49)
  4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol (NNAL) is a primary nitrosamine marker of tobacco exposure and an often-used indicator of carcinogen exposure. NNAL will be measured in urine and assessed through Liquid Chromatography-Tandem Mass Spectrometry per milligram creatinine (LC-MS/MS per mg creatinine).
Biomarkers of Exposure:1-hydroxypyrene (1-HOP) | 49 days (days 1-49)
  1-hydroxypyrene (1-HOP) is a widely used biomarker of carcinogenic polycyclic aromatic hydrocarbon exposure. 1-HOP will be measured in urine and assessed through Liquid Chromatography-Tandem Mass Spectrometry per milligram creatinine (LC-MS/MS per mg creatinine).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States